CLINICAL TRIAL: NCT02139449
Title: Prospective Study on Prognosis of Cardiac Resynchronized Therapy (CRT), Implantable Cardioverter Defibrillator (ICD) Implantation in Patients With Congestive Heart Failure (CHF)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2014-0098
Record Dates: First submitted 2014-05-13; First posted 2014-05-15 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Congestive Heart Failure
Keywords: CRT, heart failure, ICD
MeSH Terms: conditions — Heart Failure; Creatine deficiency, X-linked

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICD/CRT registry: ICD / CRTregistry in Severance or Ewha Womans University Medical Center
  Interventions: Procedure: ICD/CRT

INTERVENTIONS:
Procedure: ICD/CRT — cardiac resynchronized therapy (CRT), implantable cardioverter defibrillator (ICD) implantation

SUMMARY:
CRT and ICD has known as decreasing cardiac mortality in patient with heart failure. Especially, it has reported that CRT improved cardiac systolic function, quality of life of patients with heart failure. However, CRT and primary ICD was not generalized in Korea. So the investigators will register patients who implant CRT or ICD (primary), and follow them up. During scheduled follow up, all patients will perform echocardiography, 6 minute walking test, EKG, Holter monitoring and questionnaire on QOL.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=18
2. LV ejection fraction <40% or Clinical HF Symptom with (LV ejection fraction >40%)
3. medication for at least 3month

Exclusion Criteria:

1. patient who refuse to enroll the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with congestive heart failure(including heart failure with preserved EF or reduced EF) who are undergone cardiac resynchronized therapy (CRT), implantable cardioverter defibrillator (ICD) implantation
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-04; Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Transthoracic echocardiography (TTE) | before enrollment
Transthoracic echocardiography (TTE) | 12 month later afer enrollment
EKG | before enrollment
  for Ventricular arrhythmia events
EKG | 1 month later after enrollment
  for Ventricular arrhythmia events
EKG | 6 month later after enrollment
  for Ventricular arrhythmia events
EKG | 12 month later after enrollment
  for Ventricular arrhythmia events
NYHA(New York Heart Association) evaluation | before enrollment
  For functional capacity
  - The New York Heart Association (NYHA) Functional Classification provides a simple way of classifying the extent of heart failure. It places patients in one of four categories based on how much they are limited during physical activity; the limitations/symptoms are in regard to normal breathing and varying degrees in shortness of breath and/or angina.
NYHA(New York Heart Association) evaluation | 1 month later after enrollment
  For functional capacity
  - The New York Heart Association (NYHA) Functional Classification provides a simple way of classifying the extent of heart failure. It places patients in one of four categories based on how much they are limited during physical activity; the limitations/symptoms are in regard to normal breathing and varying degrees in shortness of breath and/or angina.
NYHA(New York Heart Association) evaluation | 6 month later after enrollment
  For functional capacity
  - The New York Heart Association (NYHA) Functional Classification provides a simple way of classifying the extent of heart failure. It places patients in one of four categories based on how much they are limited during physical activity; the limitations/symptoms are in regard to normal breathing and varying degrees in shortness of breath and/or angina.
NYHA(New York Heart Association) evaluation | 12 month later after enrollment
  For functional capacity
  - The New York Heart Association (NYHA) Functional Classification provides a simple way of classifying the extent of heart failure. It places patients in one of four categories based on how much they are limited during physical activity; the limitations/symptoms are in regard to normal breathing and varying degrees in shortness of breath and/or angina.
6 minute walking test | before enrollment
  for functional capacity
6 minute walking test | 12 month later afer enrollment
  for functional capacity

SECONDARY OUTCOMES:
Questionnaire on Quality of Life(QOL) : EQ-5D-3L (Optional) | before enrollment
  EQ-5D-3L is the scale used in the health state description part was three-level; having no problems, having some or moderate problems, being unable to do/having extreme problems. Rated level can be coded as a number 1, 2, or 3, which indicates having no problems for 1, having some problems for 2, and having extreme problems for 3. As a result, a person's health status can be defined by a 5-digit number, ranging from 11111 (having no problems in all dimensions) to 33333 (having extreme problems in all dimensions).
Questionnaire on Quality of Life(QOL) : EQ-5D-3L (Optional) | 12 month later afer enrollment
  EQ-5D-3L is the scale used in the health state description part was three-level; having no problems, having some or moderate problems, being unable to do/having extreme problems. Rated level can be coded as a number 1, 2, or 3, which indicates having no problems for 1, having some problems for 2, and having extreme problems for 3. As a result, a person's health status can be defined by a 5-digit number, ranging from 11111 (having no problems in all dimensions) to 33333 (having extreme problems in all dimensions).
Cardiac MRI or Cardiac CT | before enrollment
Cardiac MRI or Cardiac CT | 12 month later afer enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, South Korea